CLINICAL TRIAL: NCT02342652
Title: A Phase 1, Randomised, Single Blind, Placebo Controlled, 2-Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ASLAN003 in Healthy Elderly Subjects
Brief Title: A Phase 1, 2-Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ASLAN003 in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ASLAN Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ASLAN003-002
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Elderly Subjects (Age ≥55 Years)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASLAN003 (Experimental): Substance: ASLAN003 Administration route: Oral. Dosage form: Hard gelatine 50 mg capsules. Frequency: 100 mg (2 capsules) once daily for 14 consecutive days
  Interventions: Drug: ASLAN003
- Matched Placebo (Placebo Comparator): Substance: Placebo Administration route: Oral Dosage form: Hard gelatine capsules Frequency: 2 capsules once daily for 14 consecutive days
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: ASLAN003 — Healthy subject will be randomised to receive either ASLAN003 (N-aryl substituted aminoaryloic acid derivative), which is a DHODH inhibitor developed with the aim of improving several features of teriflunomide or the matching placebo as a negative control for each dose of ASLAN003 administered.
  Other Names: LAS186323
  Arms: ASLAN003
Drug: Matched Placebo — Healthy subject will be randomised to receive either ASLAN003 (N-aryl substituted aminoaryloic acid derivative), which is a DHODH inhibitor developed with the aim of improving several features of teriflunomide or the matching placebo as a negative control for each dose of ASLAN003 administered.
  Arms: Matched Placebo

SUMMARY:
This is a Phase 1, randomised, single-blind, placebo-controlled, 2 stage study design with 2 multiple dose cohorts of healthy elderly subjects.

The purpose of the study is to determine the safety, tolerability and pharmacokinetics of ASLAN003 in healthy elderly male and female subjects.

DETAILED DESCRIPTION:
This is a Phase 1, randomised, single-blind, placebo-controlled, 2 stage study design with 2 multiple dose cohorts of healthy elderly subjects.

Randomisation will be in a 3:1 ratio to ensure that 6 subjects receive ASLAN003 and 2 subjects receive placebo in a fed condition. Up to a maximum of 16 subjects (two cohorts) are planned in this study.

Subjects will be randomised to receive ASLAN003 100mg or matched placebo once daily for 14 consecutive days.

After 8 subjects have completed 14 days of dosing, the Investigator, and the Sponsor will review the available safety and PK data from all subjects before deciding to proceed with stage 2 of the study. In Stage 2, a further 8 subjects will be randomised to receive ASLAN003 100mg or matched placebo once daily for 14 consecutive days.

Following a screening visit that must fall within 28 days prior to the first dose of Investigational Product (IP) for both parts, subjects who qualify (according to the protocol-defined inclusion and exclusion criteria) will be admitted to the study centre on Day -1. Dose administration for each study part will commence on Day 1.

The subjects will stay at the study centre throughout the 14 days of dosing (D-1 toD15). Full PK blood collection will be done on D1, D8 and D14, and single trough PK blood collection on D4 and D11. All subjects will be discharged on D15 and asked to return for single PK blood sampling on D16, D17, D18, and D19 (+5days post-dose), with full outpatient visit including safety follow up and lab test on Day 19.

ELIGIBILITY:
Inclusion Criteria:

1. are capable of understanding and complying with the requirements of the study and have signed the informed consent form (ICF);
2. are able to communicate well with the Investigator, and understand and comply with the requirements of the study;
3. male or female subjects aged between 55 years and above;
4. body mass index (BMI) in the range of 18 to 27 kg/m2, inclusive;
5. healthy, as determined by pre study medical history, physical examinations, vital sign measurements, ECG (12 lead reporting RR, PR, QRS, corrected QT [QTc] using Fridericia's formulas [QTcF]) recordings with no evidence of clinically relevant medical disorders based on the opinion of the Investigator;
6. whose out-of-normal range clinical laboratory test results are not clinically relevant and are acceptable to the Investigator;
7. whose results are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening;
8. whose results are negative for drugs of abuse and alcohol tests at screening and admission to the study centre;
9. non smoker or use of < 10 cigarettes (or equivalent nicotine-containing product) per day; (able to refrain from smoking during the study period
10. male subjects must be willing to use barrier contraception during sexual intercourse, i.e. condoms, even if their partners are post-menopausal, surgically sterile or are using accepted contraceptive methods, from the first day of dose administrations until 3 months after the last dose administration;

Exclusion Criteria:

1. have participated in a study involving another investigational device or drug study within 90 days prior to randomisation in this study;
2. history of drug hypersensitivity reactions or hypersensitivity to drugs chemically related to the IP;
3. history or evidence of a clinically significant disorder, condition or disease (including, but not limited to, cardiopulmonary, oncologic, autoimmune, immunogenic, renal, metabolic, haematological or psychiatric), that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
4. existence of any surgical or medical condition which, in the judgement of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the IP;
5. clinically significant history or evidence of any active or suspected bacterial, viral, fungal or parasitic infection within the 30 days prior to randomisation (e.g. common cold, viral syndrome, flu-like symptoms, etc.);
6. active or recent history (within 30 days prior to randomisation) of acute viral infection of the skin (e.g. Herpes simplex, Molluscum contagiosum);
7. active or history of psoriasis, or a first-degree relative with active or history of psoriasis;
8. known history or evidence of active or latent tuberculosis infection (e.g. positive tuberculin skin test showing induration >5 mm or positive tuberculin blood test) in absence of previous Bacillus Calmette Guerin vaccination, or recent exposure (within 6 months prior to randomisation in this study) to an individual with active tuberculosis or with intention to travel to a country with a high risk of tuberculosis during the study period (including the follow up period);
9. history of autoimmune disease including but not limited to lupus, rheumatoid arthritis, autoimmune thyroid disease and immune thrombocytopenia;
10. QTcF values higher than 450 ms at screening, unless assessed to be non-clinically significant by the Investigator or cardiologist;
11. history of regular alcohol consumption (within 6 months prior to randomisation in this study), defined as: an average weekly intake of greater than 21 units or any average daily intake of greater than 3 units. One unit is equivalent to a half pint (220 mL) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine;
12. history of drug abuse within 1 year prior to the first day of dose administration, as judged by the Investigator and/or has a positive urine drug screen for substances of abuse including marijuana, cocaine, amphetamines, opiates, phencyclidine, barbiturates, benzodiazepines, propoxyphene, methadone metabolites, and cannabinoids and tricyclin anti-depressants at screening or on admission to the study centre;
13. has donated plasma or blood or loss of more than 250 mL blood within 1 month prior to the first day of dose administration;
14. is considering or has scheduled any surgical procedure during study participation;
15. has received any type of vaccination within 30 days prior to randomisation in this study, or is planning to receive acellular, live or attenuated vaccines during the study;
16. current use or history of use of any systemic immunomodulatory /immunosuppressive therapy, including but not restricted to systemic steroids within 3 months prior to randomisation in this study;
17. requires treatment with any medication, either prescription or non-prescription, or herbal medications, within 14 days prior to the first dose of IP (exceptions are paracetamol or vitamin products at recommended daily doses);
18. administration of any prescribed or over-the-counter drug within 2 weeks prior to screening, with the exception of paracetamol, which can be used during the study;
19. current renal insufficiency ( defined as an estimated creatinine clearance of <60 mL/min as determined from the reference range of CGH laboratory report.)
20. male subjects who plan to donate sperm in the 6 months following the receipt of IP;
21. is judged by the Investigator or the Sponsor to be inappropriate for the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety (12 lead ECGs, physical examination, vital signs measurements, pulse rate, RR, body temperature, clinical laboratory assessments and recording of adverse events) | 6 months
  Safety assessments will include 12 lead ECGs, physical examination, vital signs measurements, pulse rate, RR, body temperature, clinical laboratory assessments and recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Please contact ASLAN Pharmaceuticals, Study Director — contact@aslanpharma.com
Locations (1):
- Singapore, Singapore